CLINICAL TRIAL: NCT01650220
Title: Cardiovascular Risk Markers in Veterans With PTSD
Brief Title: Cardiovascular Risk Markers in Veterans With Post Traumatic Stress Disorder
Acronym: CVMarkers
Status: Terminated | Type: Observational
Why Stopped: The funding agency, DoD, determined that the study could not meet its enrollment numbers by the end of the grant
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: INTRuST-CV Markers
Record Dates: First submitted 2012-06-20; First posted 2012-07-26 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Disease; Post Traumatic Stress Disorder
MeSH Terms: conditions — Cardiovascular Diseases; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — For the assessment of CVD risk, high-sensitivity CRP (hs-CRP) measurements will be used. Standard assays detect 1,000 fold increases in CRP in response to infection or inflammation; these high levels cannot be used to stratify with respect to CVD risk. Hs-CRP, however, measurement can detect CRP levels as low as 0.5 mg/L. Though mainly used for research purposes, high-sensitivity IL-6 assays are also able to discriminate IL-6 levels within the normal range for CVD risk stratification. Both CRP and IL-6 levels will be analyzed as continuous quantitative traits.
  Though no DNA analysis is planned for this study, subjects are asked if they are willing to have their samples banked for future research.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Veterans with a history of PTSD
- Veterans without a history of PTSD

SUMMARY:
This is an observational study designed to determine whether veterans with PTSD have a higher risk of heart disease than those without PTSD. Cardiovascular risk will be assessed by interview and review of medical records, carotid artery ultrasound, and blood tests measuring markers of inflammation. Study participation is approximately 6 months. The eligible study population is veterans of Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), age 28 through 38 years.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF veterans at the VASDHS
* Between 28 and 38 years of age
* Willing to complete structured diagnostic interview for PTSD, CIMT ultrasound and blood test
* Willing to have a review of their medical records
* Able to give informed consent
* Have a negative urine pregnancy test, if a woman of child-bearing age

Exclusion Criteria:

* Do not meet inclusion criteria
* History of schizophrenia, other neurocognitive illness (including severe TBI by INTRuST criteria)) or active alcohol and/or drug abuse determined by chart review, interview or AUDIT-C score
* Inability to complete study tests within 18 months of study start
* Pregnancy

Ages: 28 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: OIF and OEF veterans within the VASDHS, who are between 28 and 38 years of age inclusively
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Recruitment methods feasibility | 12 months
  Comparison of the number of participants per month recruited from medical providers (with/without PTSD) vs. response to recruitment fliers (with/without PTSD) in the first 12 months of the study. Selection bias to be determined by looking at differences in age and co-morbid illnesses.
Completion of structured diagnostic interview within 2hrs. | 12 months
  Completion of Clinician Assessed PTSD Scale (CAPS), Alcohol Use Disorders Identification Test-Consumption (AUDIT-C), Patient Health Questionnaire-9 (PHQ-9), Pittsburgh Sleep Quality Index (PSQI), INTRuST Uniformed Data Set, and Family History of heart disease, within 2hrs.
Ability to schedule Carotid Intima-Media Thickness (CIMT) ultrasound in the Vascular Lab at VA San Diego Healthcare Systems, within 4 months of enrollment | 18months
  Determining whether the Vascular Lab has the capacity for a larger clinical study will be informative in planning larger prospective studies.
Time from CIMT completion to completion of clinical read. | 18months
  Rate of clinical read will help in determining adequate staffing requirements for a larger study.
Completion of serum lab measurements. | 18months

SECONDARY OUTCOMES:
Carotid Intimal Medial Thickness (CIMT) measurement | Within 4 months of subject recruitment
  CIMT thickness will be measured by carotid ultrasound
Cardiovascular Disease Biomarkers | Within 6 months of subject recruitment
  Serum C-reactive protein and interleukin-6 will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Vibha Bhatnagar, MD, Principal Investigator — University of California, San Diego
Locations (1):
- VASDHS, San Diego, California, United States